CLINICAL TRIAL: NCT03179475
Title: An Open-label, Single Centre Prospective Cohort Study to Determine the Effectiveness and Safety of Targin® for Pain Management and Opioid-induced Constipation in Patients With Spinal Cord Injury: Can we Improve Pain and Ameliorate Secondary Complications of Opioid Treatment?
Brief Title: Targin® for Chronic Pain Management in Patients With Spinal Cord Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Purdue Pharma, Canada (Industry); International Collaboration on Repair Discoveries (Other); Vancouver Coastal Health (Other Government)
Responsible Party: Principal Investigator, Andrei Krassioukov, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H16-01600
Record Dates: First submitted 2017-05-01; First posted 2017-06-07 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Chronic Pain
Keywords: Spinal Cord Injury; Traumatic Spinal Cord Injury; Targin®; Opioids; Naloxone; Opioid Induced Constipation; Oxycodone-Naloxone
MeSH Terms: conditions — Chronic Pain; Spinal Cord Injuries; Opioid-Induced Constipation | interventions — oxycodone naloxone combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oxycodone Naloxone Combination (Other): Open-Label
  Interventions: Drug: Oxycodone Naloxone Combination

INTERVENTIONS:
Drug: Oxycodone Naloxone Combination — A flexible dosing schedule will be used in this study. The dose and schedule will be based on the minimal amount of medication required to manage pain related to spinal cord injury. The dose and/or frequency will be titrated to the individual's pain level at the discretion of their regular attending physician and/or investigator.
  Oxycodone-Naloxone is available in the following oral dosages:
  1. 5 mg oxycodone hydrocholoride / 2.5 mg naloxone hydrochloride
  2. 10 mg oxycodone hydrocholoride / 5 mg naloxone hydrochloride
  3. 20 mg oxycodone hydrocholoride / 10 mg naloxone hydrochloride
  4. 40 mg oxycodone hydrocholoride / 20 mg naloxone hydrochloride
  Other Names: Targin®

SUMMARY:
The study will be investigating the effectiveness of oxycodone-naloxone (brand name Targin®) at treating chronic pain in individuals with spinal cord injury. The goal of the study is to compare the effectiveness of Targin® at treating chronic pain in individuals with sub-acute and chronic spinal cord injury compared to opioid medication that is not compounded with naloxone.

DETAILED DESCRIPTION:
This is a Phase 4, open-label prospective cohort study investigating Targin® for treating chronic pain in individuals with sub-acute and chronic spinal cord injuries. Targin® is currently approved for use by Health Canada for the treatment of moderate-to-severe chronic pain and will be investigated here for the management of moderate-to-severe chronic pain following spinal cord injury. The effectiveness and safety of opioid use for individuals with spinal cord injury has yet to be thoroughly investigated. Additionally, individuals with spinal cord injury using opioids may have the superimposed effect of neurogenic bowel and opioid induced constipation, which may cause increased frequency and severity of autonomic dysreflexia episodes, reduced quality of life, depressive symptoms, and discontinuation of opioid medication. Targin® has the potential to ameliorate these symptoms and improve treatment adherence in individuals with spinal cord injury.

ELIGIBILITY:
The inclusion criteria include, but are not limited to, the following:

* Male or female, 18 - 65 years of age
* 3 months or more following spinal cord injury
* Chronic pain for more than 3 months
* AIS score A, B, C, D with any neurological level of impairment.
* Must be taking regular opioid medication prescribed by their physician for a minimum 3 months prior to enrollment in the study
* Willing and able to comply with all clinic visits and study-related procedures
* Able to understand and complete study-related questionnaires
* Must provide informed consent

The exclusion criteria include, but are not limited to, the following:

* A daily dose of MME in excess of the maximum 120 MME (control release) or equivalent to the maximum daily dose of Targin per current Investigator Brochure or Product Monograph (80mg oxycodone hydrochloride and 40mg naloxone hydrochloride)
* Presence of severe acute medical issue that in the investigator's judgement would adversely affect the patient's participation in the study
* Imminent plan by the medical team to wean or discontinue opioid medication for pain management
* Moderate and severe forms of renal dysfunction
* Clinically significant abnormal laboratory tests as judged by the investigators.
* Hypersensitivity or allergy to opioid medication and/or naloxone.
* Use of any medication or treatment that in the opinion of the investigator indicates that it is not in the best interest of the patient to participate in this study.
* Major depression as indicated by a PHQ-9 score greater than 15 at baseline, or at the discretion of the investigator.
* Cognitive impairment as indicated by a MoCA score less than 26, or at the discretion of the investigator.
* Patient is a member of the investigational team or his/her immediate family.
* Patient does not have a good command of the English language.
* Female patients who are breast-feeding or pregnant.
* Individuals with documented substance abuse disorder
* Individuals within 1-3 months post-acute surgical intervention requiring opioid therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Change in management of pain related to spinal cord injury | 8 weeks
  Evaluation and assessment of pain is the primary objective. The evaluation tool "Revised McGill Short Form Pain" Questionnaire (SF-MPQ-2) is one of the most frequently used measures in clinical and research contexts to evaluate pain.
  The primary outcome measure is a change from baseline in SF-MPQ-2 score at 8 weeks.

SECONDARY OUTCOMES:
Change from Baseline in management of neurogenic bowel and opioid induced constipation | 8 weeks
  Evaluation and assessment of changes in neurogenic bowel and opioid-induced constipation is a secondary objective. Neurogenic bowel dysfunction, including constipation will be assessed using the evaluation tools "Neurogenic Bowel Dysfunction (NBD) score", the "Patient Assessment of Constipation-Symptoms (PAC-SYM)" score, and the "Patient Assessment of Constipation- Quality of Life (PAC-QOL)" score.
  The secondary outcome measure is a change from baseline in NBD, PAC-SYM, and PAC-QOL scores at 8 weeks.
Change from Baseline in total daily dose of medications to manage pain related to spinal cord injury | 8 weeks
  Evaluation and assessment of changes in the total daily dose of opioid medications required by individuals with spinal cord injury is a secondary objective.
  The secondary outcome measure is a change from baseline in total daily dose of opioid medications required by individuals with spinal cord injuries at 8 weeks.
Change from Baseline in total daily dose of medications to manage bowel routine | 8 weeks
  Evaluation and assessment of changes in the total daily dose of bowel routine medications required by individuals with spinal cord injury is a secondary objective.
  The secondary outcome measure is a change from baseline in the total daily dose of bowel routine medications required by individuals with spinal cord injuries at 8 weeks.
Change from Baseline of autonomic function. | 8 weeks
  Evaluation and assessment of changes in autonomic function is a secondary objective. Global autonomic function will be assessed with the neurological classification of spinal cord injury autonomic assessment form evaluation tool "International Standards on documentation of remaining Autonomic Function after Spinal Cord Injury (ISAFSCI)".
  The secondary outcome measure is a change from baseline in ISAFSCI score at 8 weeks.
Change from Baseline of quality of life. | 8 weeks
  Evaluation and assessment of changes in quality of life is a secondary objective. Quality of life will be assessed with the evaluation tool "Short Form Health Survey (SF-36)".
  The secondary outcome measure is a change from baseline in SF-36 QOL score at 8 weeks.
Change from Baseline in depressive symptoms. | 8 weeks
  Evaluation and assessment of depressive symptoms is a secondary objective. Depressive symptoms will be assessed with the evaluation tool "Patient Health Questionnaire (PHQ-9)".
  The secondary outcome measure is a change from baseline in PHQ-9 score at 8 weeks.
Change from baseline of opioid side effects. | 8 weeks
  Evaluation and assessment of opioid side effects is a secondary objective. The measure will be incidence of side effect in those treated with the study drug.
Change from baseline of opioid side effect cognitive function. | 8 weeks
  Evaluation and assessment of opioid side effects is a secondary objective. Cognitive function is of special interest to us; we will evaluate cognitive function using the evaluation tool "Montreal Cognitive Assessment (MoCA) scale".
  The secondary outcome measure is a change from baseline in MoCA score at 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Krassioukov, MD,PhD,FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Data collected during the study will be used by the investigator to communicate results of the study to the research community. Data will mostly be communicated as a pooled data set; in the event that individual participant data is communicated, it will be represented with the unique study identifier which does not identify the individual participant.